CLINICAL TRIAL: NCT05926427
Title: Orelabrutinib Combined With Rituximab and Chemotherapy for Relapsed/Refractory B-Cell Lymphoma Patients With Central Nervous System Involvement
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oreo
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: CNS Lymphoma
Keywords: CNS Lymphoma; Relapse; Refractory; orelabrutinib
MeSH Terms: conditions — Recurrence | interventions — orelabrutinib; Rituximab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OR-chemo (Experimental): Drug: Orelabrutinib, Rituximab and recommended chemotherapy according to histopathologic type
  Interventions: Drug: Orelabrutinib; Drug: Rituximab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Orelabrutinib — 150 mg qd po, until disease progression, intolerance of drug toxicity or death, otherwise maintaining during 2 years of follow-up
  Other Names: ICP-022
Drug: Rituximab — 375 mg/m^2 ivgtt, D0 of each 28-day cycle
Drug: Chemotherapy — Not specified, recommended regimen according to histopathologic type

SUMMARY:
This single-center, open, single-arm study aim to evaluate the efficacy and tolerability of a therapy introducing orelabrutinib on the basis of rituximab and chemotherapy in treating patients with relapsed or refractory B-cell lymphoma invloving central nervous system.

DETAILED DESCRIPTION:
Participants will receive orelabrutinib in addition to second-line therapy consisting of rituximab and recommended chemotherapy according to histopathologic type. After treatment of 6 cycles with the new regimen, the patients achieving CR or PR would go on to receive autologous haematopoietic stem cell transplantation (auto-HSCT) with or without orelabrutinib maintenance of 2 years (if tolerable) or orelabrutinib maintenance alone if intolerant to auto-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 80 years old;
* Histopathologically confirmed CD20 positive B-cell lymphoma according to the 5th edition of the World Health Organization (WHO) Classification of Haematolymphoid Tumours;
* After systemic treatment of the CNS lesions;
* Life expectancy of > 3 months (in the opinion of the investigator);
* No non-haematologic adverse events, except alopecia, higher than grade 1 according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0;
* Absolute Neutrophil Count (ANC) ≥ 1.0×10^9/L, Platelet Count ≥ 50×10^9/L and Haemoglobin ≥ 60 g/L, without transfusion or any use of pharmacologically hematopoietic drugs in 2 weeks;
* Serum Creatinine (SCr) ≤ 1.5 times the Upper Limit of Normal (ULN) or Creatinine Clearance Rate (CCR) ≥ 30 mL/min;
* Serum total Bilirubin (tBil) ≤ 1.5 × ULN and both Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 × ULN without hepatic metastases, otherwise tBil ≤ 3 × ULN and AST, ALT ≤ 5 × ULN respectively;
* International Normalized Ratio (INR) ≤ 1.5 and activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN;
* Left Ventricular Ejection Fraction (LVEF) ≥ 50%;
* Agreeing to provide written informed consent prior to any special examination or procedure for the research on their own or legal representative.

Exclusion Criteria:

* Pregnant or lactating women;
* Known Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infection (HBV infection refers to HBV-DNA > detectable limit);
* With acquired or congenital immunodeficiency;
* With congestive heart failure in 6 months before enrollment, New York Heart Association (NYHA) heart function class III or IV, or LVEF < 50%;
* Known to be allergic to the test drug ingredients;
* Diagnosed with or being treated for malignancy other than lymphoma;
* With severe infection;
* Substance abuse, medical, psychological, or social conditions that may interfere with the subjects' participation in the study or evaluation of the study results;
* Deemed unsuitable for the group.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | At the end-of-therapy response evaluation, 6 weeks after the end of Cycle 6, each cycle lasting 4 weeks
  The ORR is defined as percentage of participants with overall response including complete response (CR) and partial response (PR), on the basis of investigator assessments, according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
2-year Progression-Free Survival | 2 years
  Progression-free survival was defined as the time from the date of first treatment until the date of the first documented day of disease progression or relapse, according to 2014 Lugano criteria, or death from any cause, whichever occurred first.

OTHER OUTCOMES:
Overall Survival (OS) | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival is defined as the time from the date of first treatment to the date of death from any cause.
Complete Response (CR) Rate | At the end-of-therapy response evaluation, 6 weeks after the end of Cycle 6, each cycle lasting 4 weeks
  The CR rate is defined as the percentage of participants with CR, on the basis of investigator assessments, according to 2014 Lugano criteria.
Adverse Events | Baseline up to data cut-off (up to approximately 2 years)
  Any harmful reaction that occurs during the treatment of a disease according to the normal usage and dosage of a drug, which is unrelated to the purpose of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No